CLINICAL TRIAL: NCT04573400
Title: Prevalence of Neuropsychiatric Manifestations in IBD Patients in Upper Egypt
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Roshdy Abdul-Sattar, resident doctor, Assiut University
Other Study IDs: IBD and neuropsychiatry
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: IBD
MeSH Terms: interventions — 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: HADS — The HADS is a 14-item self-report questionnaire assessing levels of anxiety (seven items) and depression (seven items) over the past week. Each question is assessed on a 4-point Likert Scale: "I feel tense or 'wound up'" (0= not at all 3= most of the time). Consistent with recommendations by Bjelland et al cut-off of 8 for each HADS subscale will be used to differentiate normal from mild to severe distress.

SUMMARY:
Estimation of neuropsychiatric symptoms prevalence in IBD patients and their impact on quality of life.

DETAILED DESCRIPTION:
Crohn's disease (CD) and ulcerative colitis (UC) are the two main types of idiopathic inflammatory bowel disease (IBD), clearly distinct pathophysiological entities. UC, the most common form of IBD worldwide, is a disease of the colonic mucosa only; it is less prone to complications. In contrast, CD is a transmural disease of the gastrointestinal mucosa which can affect the entire gastrointestinal tract . CD and UC should be considered systemic diseases since they are associated with clinical manifestations involving organs outside the alimentary tract. Extraintestinal manifestations involve several organs, and either precede the onset of intestinal manifestations or appear and evolve in parallel with them . Neurologic involvement associated with IBD is frequently underreported. Nevertheless, it is important to quantify the morbidity burden of clinically significant neurologic complications in IBD because early recognition and treatment of neurologic diseases are crucial for preventing major morbidity . Neurologic involvement in IBD as a subgroup of the EIMs may precede the appearance of digestive symptoms or develop after diagnosis of IBD. In addition, neurological symptoms may exacerbate during flare-ups of IBD or evolve independently from intestinal manifestations without responding to treatment provided for the underlying bowel disease.Within (IBD) literature, anxiety and depression symptoms are commonly identified to be associated with increased disease activity and reduced quality of life. Research also indicates that ongoing psychological distress can exacerbate disease activity,] and increase the risk of flare-ups and health care costs. Given this, screening and targeted treatment of neuropsychological conditions in IBD patients are crucial.

ELIGIBILITY:
Inclusion Criteria:

* patients under the care of the hospital IBD outpatient service and having been diagnosed with IBD, aged over 18 years, and able to complete the examination and questionnaire.

Exclusion Criteria:

* Patients under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients under the care of the hospital IBD outpatient service and having been diagnosed with IBD, aged over 18 years
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Identify prevalence of neurological and psychological conditions associated with IBD. | 2021-2022

REFERENCES:
- [Background] Baumgart DC, Carding SR. Inflammatory bowel disease: cause and immunobiology. Lancet. 2007 May 12;369(9573):1627-40. doi: 10.1016/S0140-6736(07)60750-8. PMID 17499605
- [Background] Danese S, Semeraro S, Papa A, Roberto I, Scaldaferri F, Fedeli G, Gasbarrini G, Gasbarrini A. Extraintestinal manifestations in inflammatory bowel disease. World J Gastroenterol. 2005 Dec 14;11(46):7227-36. doi: 10.3748/wjg.v11.i46.7227. PMID 16437620
- [Background] Benavente L, Moris G. Neurologic disorders associated with inflammatory bowel disease. Eur J Neurol. 2011 Jan;18(1):138-43. doi: 10.1111/j.1468-1331.2010.03095.x. PMID 20500801
- [Background] Graff LA, Walker JR, Bernstein CN. Depression and anxiety in inflammatory bowel disease: a review of comorbidity and management. Inflamm Bowel Dis. 2009 Jul;15(7):1105-18. doi: 10.1002/ibd.20873. PMID 19161177
- [Background] Porcelli P, Zaka S, Centonze S, Sisto G. Psychological distress and levels of disease activity in inflammatory bowel disease. Ital J Gastroenterol. 1994 Apr;26(3):111-5. PMID 8061336
- [Background] Mittermaier C, Dejaco C, Waldhoer T, Oefferlbauer-Ernst A, Miehsler W, Beier M, Tillinger W, Gangl A, Moser G. Impact of depressive mood on relapse in patients with inflammatory bowel disease: a prospective 18-month follow-up study. Psychosom Med. 2004 Jan-Feb;66(1):79-84. doi: 10.1097/01.psy.0000106907.24881.f2. PMID 14747641
- [Background] Mardini HE, Kip KE, Wilson JW. Crohn's disease: a two-year prospective study of the association between psychological distress and disease activity. Dig Dis Sci. 2004 Mar;49(3):492-7. doi: 10.1023/b:ddas.0000020509.23162.cc. PMID 15139504